CLINICAL TRIAL: NCT00437957
Title: Phase I Trial Of Temozolomide Combined With The Histone Deacetylase Inhibitor Valproic Acid (VPA) And Whole Brain Radiation Therapy (WBR) For Brain Metastases From Solid Tumors In Adults
Brief Title: Phase I Study of Temozolomide, Valproic Acid and Radiation Therapy in Patients With Brain Metastases
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-14886; 105003A (Other: USF IRB)
Record Dates: First submitted 2007-02-19; First posted 2007-02-21 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2011-06

CONDITIONS: Brain Metastases
Keywords: histone deacetylase; unresectable brain metastases
MeSH Terms: conditions — Brain Neoplasms | interventions — Temozolomide; Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Temazolomide, Valproic Acid and Radiation (Experimental): Temazolomide, Valproic Acid and Whole Brain Radiation Therapy
  Interventions: Drug: Temozolomide; Drug: Valproic Acid; Procedure: Whole Brain Radiation Therapy

INTERVENTIONS:
Drug: Temozolomide — 75 Mg/m2/day for all Cohorts
  Other Names: Temodar
Drug: Valproic Acid — Cohort 1: 20 mg/kg/day Cohort 2: 30 mg/kg/day Cohort 3: 40 mg/kg/day Cohort 4: 50 mg/kg/day
  Other Names: VPA
Procedure: Whole Brain Radiation Therapy — Concurrently with Temozolomide and VPA
  Other Names: WBRT

SUMMARY:
This type of study is called a "Phase I study". Its purpose is to determine the side effects of the two medicines listed in this study when given together with whole brain radiation, and the highest dose of valproic acid that can be given together with temozolomide and whole brain radiation. We will also study the drug combination's effectiveness in treating cancer. While both of these drugs and whole brain radiation have been used in people for many years, they have never been combined for the purpose of treating patients with cancer.

DETAILED DESCRIPTION:
At the start of the study, patients will be informed which dose level they will be treated with. On day 1, patients will have a physical exam and several blood draws including draws to measure the level of valproic acid in their body. Patients will start your whole brain radiation and also at the same time start the valproic acid and temozolomide pills. Patients will be asked to take the valproic acid pills every 12 hours and the temozolomide pills once daily. Patients will not need to come to the center for that but will need to come to the center to receive you whole brain radiation for 3 weeks (on weekdays, excluding holidays). Radiation therapy will not be administered on weekends but patients will still take their pills for the whole 3 weeks from starting the radiation.

Patients will have to come back for a study visit weekly for the 6 months. Two more visits are also required: approximately 6 weeks and 10 weeks from starting the treatment. Patients will be asked about any old or new symptoms to determine if adjustment in the pill dose is required.

Every study visit except the last one will include blood draws. These will evaluate blood counts, blood chemistry and also measure the level of valproic acid in your body. The Mini Mental Status examination described above will be repeated in every visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have cytologically/histologically documented solid tumor malignancies
* Age > 18 years old
* Patients must be candidates to receive WBR for unresectable brain metastases
* Patients must have ECOG performance status 0-2
* Patients must be able to give informed consent and able to follow guidelines given in the study
* Neurologic Function Status 0,1, or 2
* The patient has no major impairment of hematological function, as defined by the following laboratory parameters: WBC >3.0x10^9/L; ANC > 1.5 x 10^9/L; Hgb >9.0g/dL; PLT >100x10^9/L. Red blood cell transfusions and repeat evaluations for study entry are allowed
* Patients must have adequate renal and normal hepatic function (creatinine < 1.5 x upper limit of normal (ULN), bilirubin and SGOT (AST), SGPT (ALT) within 1.5 x the upper institutional normal limits) obtained within 4 weeks prior to registration.
* All patients of reproductive potential must use an effective method of contraception during the study and six months following termination of treatment. (Not applicable to patients with bilateral oophorectomy and/or hysterectomy or to female patients who are older than 50 years and have not had a menstrual cycle in more than one year).
* Women of childbearing age must have a negative pregnancy test
* Patients must have 10 mm or greater brain lesion on MRI scan performed within 4 weeks of enrollment

Exclusion Criteria:

* Prior whole brain radiation
* More than 1 active malignancy which may potentially cause brain metastasis
* Patients on phenytoin, carbamazepine, phenobarbital, felbamate, meropenem, rifampin (Levetiracetam will be permitted)
* Patients with active or any history of seizure disorders
* Patients with uncontrolled nausea and vomiting
* Chemotherapy, radiotherapy, or hormonal therapy within 2 weeks prior to entering the study or have not recovered from prior treatment-related toxicities (grade 2 or less)
* Patients receiving any other investigational agents
* Evidence of significant active infection (e.g., pneumonia, cellulitis, wound abscess, etc.) at time of study entry.
* Leptomeningeal disease or hydrocephalous on MRI scan performed within 4 weeks of enrollment
* Pregnant and breast feeding women are excluded from the study because effects on the fetus are unknown and there may be a risk of increased fetal wastage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-12; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of temozolomide in combination with VPA and Whole-Brain Radiation | approximately 74 days per patient
Determination of the MTD of VPA in combination with temozolomide and Whole-Brain Radiation | approximately 74 days per patient

SECONDARY OUTCOMES:
Response rate | approximately 74 days per patient
Pharmacokinetics | approximately 74 days per patient
Histone acetylation | approximately 74 days per patient

CONTACTS AND LOCATIONS:
Overall Officials: Sajeel Chowdhary, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute; Jade Homsi, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States